CLINICAL TRIAL: NCT03500744
Title: Erector Spinae Plane Block for Major Gynecologic and Urologic Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit due to COVID situation and protocols
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Kamal Kumar, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111510
Record Dates: First submitted 2018-03-17; First posted 2018-04-18 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Hysterectomy; Cystectomy; Regional Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Sham block will be performed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector spinae plane block (Experimental): The ESPB will be performed with ultrasound guidance. After identifying a suitable location between 8th and 10th thoracic spine transverse process, the overlying skin will be infiltrated with local anesthetic. A 22 gauge 90-mm needle will be inserted to make contact with the transverse process and withdraw slightly. Ropivacaine 0.5% 20 mL will be injected at this location. The same procedure will be performed on the other side.
  Additionally, patients will receive acetaminophen, gabapentin and intravenous patient-controlled analgesia opioids.
  Interventions: Procedure: Erector spinae plane block
- Shame block (Sham Comparator): A sham block will be performed by performing ultrasound examination of the back looking for intended location for ESPB placement. Skin will be infiltrated with local anesthetics but ESPB will not be performed.
  Additionally, patients will receive acetaminophen, gabapentin and intravenous patient-controlled analgesia opioids.
  Interventions: Procedure: Sham block

INTERVENTIONS:
Procedure: Erector spinae plane block — Ropivacaine 0.5% 20 mL at each site of ESPB
  Arms: Erector spinae plane block
Procedure: Sham block — Skin infiltration only
  Arms: Shame block

SUMMARY:
Regional anesthesia, also know as a nerve block, is a key component of pain control after major abdominal surgery. Bilateral erector spinae plane block (ESPB) performed at low thoracic level has been shown to be an effective pain control method in case reports. This pilot study aims to further characterize the pain-control characteristics and to provide baseline data for future trials.

ELIGIBILITY:
Inclusion Criteria:

Adult surgical patients who are American Society of Anesthesiologists (ASA) class I to III, undergoing cystectomy, or total abdominal hysterectomy, salpingo-oophrectomy with or without omentectomy via midline laparotomy.

Exclusion Criteria:

1. BMI > 40
2. Non-English speaking
3. Patient refusal or inability to consent
4. Cognitive or psychiatric history that would make it difficult to assess pain score
5. Pre-existing chronic pain condition
6. Preoperative opioid use greater than the equivalent of oral morphine 30 mg daily
7. Infection over site of block placement
8. Allergy or contraindication to any study medication
9. Coagulopathy or thrombocytopenia
10. Postoperative ICU admission
11. Presence of significant cardiac, respiratory, hepatic, renal or neurologic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | First 12 postoperative hour
  Postoperative opioid consumption in oral morphine equivalents
Pain score | First 12 postoperative hour
  Numeric rating scale (0 - 10) for pain score, area under curve first 12 hours

SECONDARY OUTCOMES:
Length of stay in post-anesthetic recovery unit | until discharge from post-anesthetic recovery unit, up to 4 hours postoperaively
  Length of stay in post-anesthetic recovery unit
Length of stay in hospital | until discharge from hospital, up to 7 days postoperatively
  Length of stay in hospital
Number of participants with opioid related complication | Until discharge, up to 7 days postoperatively
  Nausea, vomiting, pruritus
Number of participants with block related complication | Until discharge, up to 7 days postoperatively
  Hematoma, nerve deficit, pneumothorax
Pain score 12 - 24 hour | 12th to 24th postoperative hour
  Area under curve of Numeric rating scale(0 - 10) pain score during the 12 to 24th postoperative hour
Opioid consumption 12 - 24 hour | 12th to 24th postoperative hour
  Postoperative opioid consumption in oral morphine equivalents

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Lin, Principal Investigator — Western University
Locations (1):
- Cheng Lin, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided